CLINICAL TRIAL: NCT00227448
Title: Induced Hypertension for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01-NS-042607-1; R01NS042607 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Ischemic; Stroke
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke | interventions — Midodrine

INTERVENTIONS:
Drug: intravenous saline
Drug: intravenous phenylephrine
Drug: intravenous levophed
Drug: oral midodrine

SUMMARY:
The ultimate goal of this multicenter, phase II study is to increase blood pressure until either a neurologic response is seen or a target mean arterial pressure of 30% above baseline is achieved. IV fluids, IV phenylephrine and/or IV norepinephrine are used to rapidly raise mean arterial pressure in a controlled manner as serial assessments of neurologic function are performed.

DETAILED DESCRIPTION:
This is a multicenter, pilot clinical trial. The primary outcome variables will be the presence or absence of improvement in NIHSS during treatment with induced hypertension and the number of adverse events. The secondary outcome variables will be final infarct size on MRI at 1 month and Barthel Index and Modified Rankin Scale at 3 months.

All patients fulfilling the inclusion and exclusion criteria and who are willing to participate will receive intervention to induce hypertension, including intravenous saline, phenylephrine (neosynephrine) or levophed, and possibly oral midodrine. Blood pressure will be increased to a maximum mean arterial pressure (MAP) that is 30% above the baseline MAP as measured in the emergency department. The acute phase of the study will last for 3-5 days (for responders) and all patients will be followed up at 1 and 3 months post stroke onset. All patients will undergo neurologic, cognitive, and physical examinations as well as serial MRI studies with diffusion and perfusion-weighted imaging.

Primary hypotheses will be measured using the National Institutes of Health Stroke Scale (NIHSS) and MRI. Improvement following induced hypertension will be measured by comparing NIHSS performed at multiple time points throughout the study. The ability to predict diffusion-perfusion mismatch will be determined by comparing MRI #1 and MRI #2. NIHSS and MRI will also be compared to determine if NIHSS correlates with reperfusion area on MRI.

The secondary hypothesis of improved long-term outcome will be measured using the Barthel Index, the modified Rankin Scale, and MRI/Flair at 1 and 3 months post stroke symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke in whom treatment can be initiated within 12 hours of a clearly defined symptom onset. (If the patient awakens with a deficit, time of onset is considered the time the patient was last seen functioning normally.)
* Age older then 18 years of age.
* Measurable neurologic deficit other than isolated facial weakness, sensory loss or ataxia. NIHSS must be > 4 points.
* Head CT showing no evidence of intracranial hemorrhage or mass lesion which might increase the risk of bleeding.
* Absence of ischemic changes on EKG (i.e. > than 1mm ST segment elevation or depression in at least two contiguous leads, new T waves inversion in two leads).
* No contraindication to MRI studies, including allergy to gadolinium.

Exclusion Criteria:

* History of unstable angina, any recent angina (defined as chest pain) in the past 3 months, recent myocardial infarction (less then 3 months), any history of ventricular arrhythmia, presence of left ventricular bundle branch block on EKG.
* History of severe and symptomatic cardiac valvular disease.
* History of congestive heart failure, dilated cardiomyopathy, hypertrophic obstructive cardiomyopathy, or known ejection fraction < 25%.
* Systolic blood pressure greater > 200 mm Hg or MAP > 120 mm HG when patient is initially monitored.
* Serum creatinine greater then 2 mg/dl.
* History of symptomatic peripheral vascular disease or Raynaud's syndrome.
* Suspected seizure at the onset of stroke.
* Treatment with IV tPA or other thrombolytic agent.
* Massive stroke (> 2/3 MCA territory) or any amount of midline shift due to cerebral edema on head CT.
* Pregnancy
* Current use of MAO inhibitors, tricyclic antidepressant medications, or cyclopropane or halothane anesthetic agents.
* Coma.
* Allergies or known contraindications to the use of IV phenylephrine, IV norepinephrine, sodium metabisulfite, or oral midodrine.
* Hemorrhage on initial MRI or CT or other structural lesion that might raise the risk of intracranial bleeding.
* Thrombocytopenia (plt < 100 k), PTT > 100 sec, INR > 3.0 at time of treatment.
* Participation in other investigational trial within 30 days.
* Moderate to severe baseline disability (pre-stroke Rankin score of > 3), severe or terminal concurrent medical illness with expected survival of < 3 months, or other concurrent medical or psychiatric condition which may limit neurologic assessment or patient follow-up in the opinion of the investigator.
* Requirement for anticoagulation with IV heparin or warfarin in the first 48 hours after enrollment.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
* Toxicology screen positive for cocaine.
* Intubated at time of enrollment.
* Mesenteric or peripheral vascular thrombosis.
* Profound hypoxia or hypercarbia as defined as a PaO2 level less than 50 or a PaCO2 level of greater than 60.
* Norepinephrine Exclusion Criteria- The patient will not receive Norepinephrine if the patient has any of the following: lack of sufficient vascular access (central line or peripheral line greater than 18 gauge is sufficient), hypersensitivity to norepinephrine products, severe hypertension as in 4.2.4 above, tachycardia defined as HR >100 for 10 minutes sustained, myocardial infarction, pulmonary edema, peripheral ischemia, or ventricular arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-06; Study Completion 2005-04

PRIMARY OUTCOMES:
NIHSS during the intervention and at 30 and 90 days
MRI at post intervention

SECONDARY OUTCOMES:
Barthel Index at 30 and 90 days
Rankin at 30 and 90 days
MRI at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wityk, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts